CLINICAL TRIAL: NCT02722304
Title: A Stage 1, Prospective, Randomized, Placebo-Controlled, Double- Blind Study to Evaluate the Safety and Efficacy of Alpha1-Proteinase Inhibitor (A1PI) Augmentation Therapy in Subjects With A1PI Deficiency and Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Stage 1 Study of ARALAST NP and GLASSIA in A1PI Deficiency
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 460503
Record Dates: First submitted 2016-03-23; First posted 2016-03-30 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Alpha1-antitrypsin Deficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (5):
- ARALAST NP 60 mg/kg (Experimental): 60 mg/kg body weight/week
  Interventions: Biological: ARALAST NP 60 mg/kg
- ARALAST NP 120 mg/kg (Experimental): 120 mg/kg body weight/week
  Interventions: Biological: ARALAST NP 120 mg/kg
- GLASSIA 60 mg/kg (Experimental): 60 mg/kg body weight/week
  Interventions: Biological: GLASSIA 60 mg/kg
- GLASSIA 120 mg/kg (Experimental): 120 mg/kg body weight/week
  Interventions: Biological: GLASSIA 120 mg/kg
- Placebo (Placebo Comparator): Human Albumin 2%
  Interventions: Biological: Human Albumin 2%

INTERVENTIONS:
Biological: ARALAST NP 60 mg/kg — ARALAST NP is an Alpha1-Proteinase Inhibitor (A1PI) augmentation therapy
  Other Names: Alpha1-Proteinase Inhibitor (Human); A1PI; Alpha1-Proteinase Inhibitor
  Arms: ARALAST NP 60 mg/kg
Biological: ARALAST NP 120 mg/kg — ARALAST NP is an Alpha1-Proteinase Inhibitor (A1PI) augmentation therapy
  Other Names: Alpha1-Proteinase Inhibitor; Alpha1-Proteinase Inhibitor (Human); A1PI
  Arms: ARALAST NP 120 mg/kg
Biological: GLASSIA 60 mg/kg — GLASSIA is an Alpha1-Proteinase Inhibitor (A1PI) augmentation therapy
  Other Names: Alpha1-Proteinase Inhibitor (Human); A1PI; Alpha1-Proteinase Inhibitor
  Arms: GLASSIA 60 mg/kg
Biological: GLASSIA 120 mg/kg — GLASSIA is an Alpha1-Proteinase Inhibitor (A1PI) augmentation therapy
  Other Names: Alpha1-Proteinase Inhibitor; Alpha1-Proteinase Inhibitor (Human); A1PI
  Arms: GLASSIA 120 mg/kg
Biological: Human Albumin 2% — Human albumin 2% (by appropriate dilution with normal saline solution)
  Arms: Placebo

SUMMARY:
The purpose of this study is to conduct a pilot study to evaluate the safety and efficacy of weekly administration of Alpha1-Proteinase Inhibitor (A1PI) augmentation therapy in subjects with A1PI deficiency and emphysema/ chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at the time of screening
2. Endogenous plasma Alpha1-Proteinase Inhibitor (A1PI) level <8 μM at any time during the Screening period for treatment-naïve participants, or following 4-weeks minimum wash-out from previous augmentation therapy in treatment-experienced participants. The screening plasma A1PI level may be repeated if a participant obtains an exclusionary value that is suspected to be due to inadequate washout of A1PI).
3. Participant has documented A1PI genotype of Pi*Z/Z, Pi*Z/Null, Pi*Malton/Z, Pi*Null/Null, or other rare genotypes (except PI*MS, PI*MZ, or PI*SZ).
4. Clinically evident mild-moderate chronic obstructive pulmonary disease (COPD) (according to GOLD criteria for diagnosis) at the time of screening.
5. If the participant is treated with any respiratory medications including inhaled bronchodilators, inhaled corticosteroids, or systemic corticosteroids (e.g. prednisone ≤ 10 mg/day or its equivalent), the doses of the participant's medications have remained stable for at least 28 days prior to screening.
6. No clinically significant abnormalities (other than emphysema, bronchitis or bronchiectasis) detected via a chest computed tomography (CT) or chest X-ray at the time of screening.
7. If female of childbearing potential, participant must have a negative pregnancy test at screening and agree to employ adequate birth control measures for the duration of the study.
8. Participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Known ongoing or history of clinically significant pulmonary impairment other than emphysema/ COPD.
2. The participant is experiencing lower respiratory infection (LRTI)/acute pulmonary exacerbation (APE) at the time of enrollment (signing Informed consent form (ICF)). Participant may be rescreened after both clinical resolution of LRTI/APE and having also remained stable for at least 4 weeks after the end of LRTI/APE).
3. Known ongoing or history of cor pulmonale.
4. Known resting partial pressure of carbon dioxide (PaCO2) levels of > 45 mmHg.
5. Clinically significant congestive heart failure with New York Heart Association (NYHA) Class III/IV symptoms.
6. The participant has received an organ transplant, has undergone major lung surgery, or is currently on a transplant list.
7. Known history of ongoing malignancy (other than adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix).
8. Smoker or participant that has ceased smoking for less than one year prior to screening whose levels of cotinine are outside of the normal range of a nonsmoker.

   All participants must agree to refrain from smoking throughout the course of the study.
9. The participant is receiving long-term therapy (> 28 days) of parenteral corticosteroids or oral corticosteroids at doses greater than 10 mg/day of prednisone or its equivalent).
10. The participant is receiving long-term round-the-clock oxygen supplementation (other than temporary for acute COPD exacerbation, or supplemental oxygen (O2) with continuous positive airway pressure [CPAP], or bi-level positive airway pressure [BiPAP] during the day).
11. Participant has contraindications for CT (e.g. body weight and/or body size exceeding the weight and gantry size limits specified by the manufacturer of the CT scanner, inability to lie flat in the CT scanner, claustrophobia, metal prosthesis or pacemaker in the chest wall or upper extremity that would impact lung density assessment).
12. Participant is unwilling or unable to modify bronchodilator medications for 6 hours for short acting β2 agonists, 24 hours for long-acting β2 agonists, and 48 hours for long acting anticholinergics prior to the scheduled quantitative CT scan.
13. Known severe immunoglobulin A (IgA) deficiency (ie, IgA level < 8 mg/dL at screening).
14. Known history of hypersensitivity following infusions of human blood or blood components (eg, human immunoglobulins or human albumin).
15. Presence of clinically significant laboratory abnormalities at the screening
16. The participant has a clinically significant medical, psychiatric, or cognitive illness, is a recreational drug/alcohol user, or has any other uncontrolled medical condition (eg, unstable angina, transient ischemic attack, uncontrolled hypertension) that, in the opinion of the investigator, would affect participant's safety or compliance or confound the results of the study.
17. Participant has been exposed to another IP within 28 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
18. Participant is a family member or employee of the investigator.
19. If female, participant is pregnant or nursing at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (17):
- United States (14):
  - Phoenix Medical Research Institute, LLC, Peoria, Arizona
  - Newport Native MD, Inc, Newport Beach, California
  - Pulmonary Disease Specialists, P.A., / PDS Research, Kissimmee, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - Loyola University Health System, Maywood, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - La Porte County Institute for Clinical Research, Inc., Michigan City, Indiana
  - Pulmonary Health Physicians, Fayetteville, New York
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Southeastern Research Center LLC, Winston-Salem, North Carolina
  - Metroplex Pulmonary and Sleep Center, Allen, Texas
  - Houston Pulmonary and Sleep Associates, Houston, Texas
  - Element Research Group, San Antonio, Texas
  - Renovatio Clinical-Respiratory & Sleep Disorders Specialists, The Woodlands, Texas
- St Vincent's Hospital Melbourne, Fitzroy, Victoria, Australia
- Canada (2):
  - LHSC - Victoria Hospital, London, Ontario
  - Inspiration Research Limited, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 study centers in the United States (3) and Australia (1) between 02 November 2016 (first participant first visit) and 14 September 2018 (last participant last visit).
Pre-assignment Details: A total of 22 participants were screened for entry of study, of these, 15 participants were considered screen failures. Remaining 7 participants were enrolled and randomized in the study.
Groups:
- ARALAST NP 60 mg/kg (Group 1): Participants received 60 milligram per kilogram body weight per week (mg/kg BW/week) of ARALAST NP intravenous (IV) infusion for a total of 96 weeks.
- ARALAST NP 120 mg/kg (Group 2): Participants received 120 mg/kg BW/week of ARALAST NP IV infusion for a total of 96 weeks.
- GLASSIA 60 mg/kg (Group 3): Participants received 60 mg/kg BW/week of GLASSIA IV infusion for a total of 96 weeks.
- GLASSIA 120 mg/kg (Group 4): Participants received 120 mg/kg BW/week of GLASSIA IV infusion for a total of 96 weeks.
- Placebo (Group 5): Participants received 6 milliliter per kilogram body weight per week (ml/kg BW/week) of placebo (human albumin two percent [%]) in normal saline for a total of 96 weeks.
Period: Overall Study
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | ARALAST NP 120 mg/kg (Group 2) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5)
Started | 1 | 0 | 2 | 2 | 2
Treated | 1 | 0 | 1 | 1 | 2
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 2 | 2 | 2
Not completed — Study Terminated by Sponsor | 1 | 0 | 2 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all participants who had received any amount of investigational product (IP) or placebo, regardless of protocol deviations or non-adherence to the study procedures. Analysis was performed according to the treatment regimen received regardless of the randomized treatment regimen.
Groups:
- Total: Total of all reporting groups
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | ARALAST NP 120 mg/kg (Group 2) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5) | Total
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (NA) — Standard Deviation was not calculated as only one participant was evaluated. |  | 65.0 (NA) — Standard Deviation was not calculated as only one participant was evaluated. | 68.0 (NA) — Standard Deviation was not calculated as only one participant was evaluated. | 46.0 (4.24) | 57.4 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1 | 1 | 2 | 5
  Male | 0 |  | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 |  | 1 | 1 | 2 | 5
  Unknown or Not Reported | 0 |  | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0 | 0 | 0
  Asian | 0 |  | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0 | 0 | 0
  Black or African American | 0 |  | 0 | 0 | 0 | 0
  White | 1 |  | 1 | 1 | 2 | 5
  More than one race | 0 |  | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change in Lung Density Based on Group 1 (ARALAST NP) Versus Placebo, Group 3 and Group 4 (GLASSIA) Versus Placebo
Description: Rate of change in lung density was assessed by computed tomography (CT) densitometry. Computed Tomography (CT) scans was used to measure lung density as a quantitative assessment of emphysema progression and treatment efficacy at each of the study visits. CT lung density at the 15th percentile (PD15) is the threshold below which 15% of the voxels have lower densities, and was used as the parameter for estimating the rate of lung density decline. Rate of change in lung density based on Group 1 (ARALAST NP) versus Placebo, Group 3 and Group 4 (GLASSIA) versus Placebo were reported. The safety analysis set used for all the efficacy parameter assessment.
Time Frame: Baseline, Early termination of the study (approximately 22 months)
Population: Study was early terminated due to low and slow rate of enrollment, hence, data was not collected for this efficacy endpoint.
Groups:
- ARALAST NP 60 mg/kg Versus Placebo: Participants received 60 milligram per kilogram body weight per week (mg/kg BW/week) of ARALAST NP intravenous (IV) infusion and 6 milliliter per kilogram body weight per week (ml/kg BW/week) of placebo (human albumin two percent [%]) in normal saline for a total of 96 weeks.
- GLASSIA 60 mg/kg Versus Placebo: Participants received 60 mg/kg BW/week of GLASSIA IV infusion and 6 ml/kg BW/week of placebo (human albumin two %) in normal saline for a total of 96 weeks.
- GLASSIA 120 mg/kg Versus Placebo: Participants received 120 mg/kg BW/week of GLASSIA IV infusion and 6 ml/kg BW/week of placebo (human albumin two %) in normal saline for a total of 96 weeks.
Arm/Group | ARALAST NP 60 mg/kg Versus Placebo | GLASSIA 60 mg/kg Versus Placebo | GLASSIA 120 mg/kg Versus Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Rate of Change in Lung Density for Each Treatment Group
Description: Rate of change in lung density was assessed by computed tomography (CT) densitometry for each treatment group. Computed Tomography (CT) scans was used to measure lung density as a quantitative assessment of emphysema progression and treatment efficacy at each of the study visits. The safety analysis set used for all the efficacy parameter assessment.
Time Frame: Baseline, Early termination of the study (approximately 22 months)
Population: as for outcome 1
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5)
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Mean Steady State Trough Concentration of Antigenic and Functional Alpha1-Proteinase Inhibitor (A1PI) for ARALAST NP and GLASSIA at Each Dose Level
Description: Mean steady state trough concentration of antigenic and functional alpha1-proteinase inhibitor (a1pi) for ARALAST NP and GLASSIA at each dose level was reported.
Time Frame: Baseline, Early termination of the study (approximately 22 months)
Population: as for outcome 1
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5)
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Events With Related and Unrelated Serious and Non-Serious Treatment Emergent Adverse Event (TEAE)
Description: An Adverse event (AE) was defined as any untoward medical occurrence in a participant administered an IP that does not necessarily have a causal relationship with the treatment. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were defined as AEs with a start date on or after the first dose of double-blind investigational product or a start date before the date of the first dose of double-blind investigational product that increased in severity or after the date of the first dose. TEAE related to Investigational Product (IP) and Study Procedures (SP) were considered. A non-serious AE is an AE that does not meet the criteria of an SAE. Number of events with related and unrelated serious and non-serious TEAE were reported.
Time Frame: From start of study treatment up to early termination of the study (approximately 22 months)
Population: SAS included all participants who had received any amount of IP or placebo, regardless of protocol deviations or non-adherence to the study procedures. Analysis was performed according to the treatment regimen received regardless of the randomized treatment regimen.
Measure: Number; unit: Events
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5)
Number analyzed (Participants) | 1 | 1 | 1 | 2
Events
  Serious TEAE: Events Related to IP | 0 | 0 | 0 | 0
  Non-serious TEAE: Events Related to IP | 0 | 0 | 0 | 19
  Serious TEAE: Events Related to SP | 0 | 0 | 0 | 0
  Non-serious TEAE: Events Related to SP | 0 | 0 | 0 | 1
  Serious TEAE: Unrelated Events | 0 | 0 | 0 | 0
  Non-serious TEAE: Unrelated Events | 2 | 0 | 0 | 5

5. Secondary Outcome: Percentage of Participants With Related and Unrelated Serious and Non-Serious Treatment Emergent Adverse Events (TEAE's)
Description: An Adverse event (AE) was defined as any untoward medical occurrence in a participant administered an IP that does not necessarily have a causal relationship with the treatment. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were defined as AEs with a start date on or after the first dose of double-blind investigational product or a start date before the date of the first dose of double-blind investigational product that increased in severity or after the date of the first dose. A non-serious AE is an AE that does not meet the criteria of an SAE. TEAE related to IP and Study Procedures were considered. Percentage of participants with related and unrelated serious and non-serious TEAE were reported.
Time Frame: From start of study treatment up to early termination of the study (approximately 22 months)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5)
Number analyzed (Participants) | 1 | 1 | 1 | 2
Percentage of Participants
  Serious TEAE: Related to IP | 0 | 0 | 0 | 0
  Non-Serious TEAE: Related to IP | 0 | 0 | 0 | 50
  Serious TEAE: Related to SP | 0 | 0 | 0 | 0
  Non-Serious TEAE: Related to SP | 0 | 0 | 0 | 50
  Serious TEAE: Unrelated | 0 | 0 | 0 | 0
  Non-Serious TEAE: Unrelated | 100 | 0 | 0 | 100

6. Secondary Outcome: Number of Events With Temporally Related Serious and Non-Serious Treatment Emergent Adverse Events (AEs)
Description: An Adverse event (AE) was defined as any untoward medical occurrence in a participant administered an IP that does not necessarily have a causal relationship with the treatment. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were defined as AEs with a start date on or after the first dose of double-blind investigational product or a start date before the date of the first dose of double-blind investigational product that increased in severity or after the date of the first dose. A non-serious AE is an AE that does not meet the criteria of an SAE. TEAEs were temporally related to treatment administration (ie, occurred within 72 hours following the end of the infusion). TEAE Related to IP were considered.
Time Frame: From start of study treatment up to early termination of the study (approximately 22 months)
Population: SAS included all participants who had received any amount of IP or placebo, regardless of protocol deviations or non-adherence to the study procedures. Analysis was performed according to the treatment regimen received regardless of the ( randomized treatment regimen.
Measure: Number; unit: Events
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5)
Number analyzed (Participants) | 1 | 1 | 1 | 2
Events
  Temporally Serious TEAE Related to IP | 0 | 0 | 0 | 0
  Temporally Non-Serious TEAE Related to IP | 0 | 0 | 0 | 17

7. Secondary Outcome: Percentage of Participants With Temporally Related Serious and Non-Serious Treatment Emergent Adverse Events (AEs)
Description: as for outcome 6
Time Frame: From start of study treatment up to early termination of the study (approximately 22 months)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5)
Number analyzed (Participants) | 1 | 1 | 1 | 2
Percentage of Participants
  Temporally Serious TEAE Related to IP | 0 | 0 | 0 | 0
  Temporally Non-Serious TEAE Related to IP | 0 | 0 | 0 | 50

8. Secondary Outcome: Number of Events With Suspected Adverse Reactions or Serious and Non-Serious Adverse Reactions (ARs)
Description: An Adverse Reactions (ARs) plus suspected adverse reaction is any adverse event which met any of the following criteria: an adverse event that began during infusion or within 72 hours following the end of IP infusion; an adverse event considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration; an adverse event for which causality assessment was missing or indeterminate. Adverse reaction included both serious and non-serious ARs.
Time Frame: From start of study treatment up to early termination of the study (approximately 22 months)
Population: SAS included all participants who had received any amount of investigational product (IP) or placebo, regardless of protocol deviations or non-adherence to the study procedures. Analysis was performed according to the treatment regimen received regardless of the randomized treatment regimen.
Measure: Number; unit: Events
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5)
Number analyzed (Participants) | 1 | 1 | 1 | 2
Events
  Suspected ARs or Non-serious ARs | 1 | 0 | 0 | 24
  Suspected ARs or Serious ARs | 0 | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants With Suspected Adverse Reactions or Serious and Non-Serious Adverse Reactions (ARs)
Description: An Adverse Reactions (AR) plus suspected adverse reaction is any adverse event which met any of the following criteria: an adverse event that began during infusion or within 72 hours following the end of IP infusion; an adverse event considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration; an adverse event for which causality assessment was missing or indeterminate. Adverse reaction included both serious and non-serious ARs.
Time Frame: From start of study treatment up to early termination of the study (approximately 22 months)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5)
Number analyzed (Participants) | 1 | 1 | 1 | 2
Percentage of Participants
  Suspected ARs or Non-serious ARs | 100 | 0 | 0 | 50
  Suspected ARs or Serious ARs | 0 | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants With at Least One Infusion Rate Change or Infusion Interruption or Stopped Due to AEs
Description: An Adverse event (AE) was defined as any untoward medical occurrence in a participant administered an IP that does not necessarily have a causal relationship with the treatment. Number of infusions for which the infusion rate was reduced and/or the infusion interrupted or stopped due to adverse events (AEs) were reported.
Time Frame: From start of study treatment up to early termination of the study (approximately 22 months)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5)
Number analyzed (Participants) | 1 | 1 | 1 | 2
Percentage of Participants
  Participants with at Least 1 Infusion Rate Change | 0 | 0 | 0 | 50
  Participantswith at Least 1 Infusion Interruption | 0 | 0 | 0 | 50

11. Secondary Outcome: Number of Participants Who Developed Anti-A1PI Antibodies Following Treatment With ARALAST NP or GLASSIA
Description: Number of participants who developed anti- A1PI antibodies following treatment with ARALAST NP or GLASSIA were reported. Anti-A1PI binding antibody were determined for the samples that tested positive or negative at each assessment time point.
Time Frame: Baseline, Early termination of the study (approximately 22 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5)
Number analyzed (Participants) | 1 | 1 | 1 | 2
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment up to early termination of the study (approximately 22 months)
Description: Study was terminated early. One arm/ group (ARALAST NP 120 mg/kg (Group 2)) did not have any participants randomized to it at the time of the study termination. Therefore there are zero participants at risk. This applies to the following fields, below for the ARALAST NP 120 mg/kg (Group 2) arm/group: - participants at risk for Serious Adverse Events - participants at risk for All-Cause Mortality - participants at risk for Other (Not Including Serious) Adverse Events
Arm/Group | ARALAST NP 60 mg/kg (Group 1) | ARALAST NP 120 mg/kg (Group 2) | GLASSIA 60 mg/kg (Group 3) | GLASSIA 120 mg/kg (Group 4) | Placebo (Group 5)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/1 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/1 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/1 | 0/1 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARALAST NP 60 mg/kg (Group 1) (N=1) | ARALAST NP 120 mg/kg (Group 2) (N=0) | GLASSIA 60 mg/kg (Group 3) (N=1) | GLASSIA 120 mg/kg (Group 4) (N=1) | Placebo (Group 5) (N=2)
Right Eye Retinal Detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13)
Nausea (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
CONTACT DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
site conditions/ Catheter site rash/ MILD RASH AT THE SITE OF TAPE USED AT IV CANNULA SITE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage/ PER VAGINAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Chronic obstructive pulmonary disease/ COPD EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The Data Monitoring Committee (DMC) reviewed the available efficacy and safety data and unanimously recommended to terminate the study. The decision was based on the very low number of enrollees, and the slow rate of participant enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT02722304/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT02722304/SAP_001.pdf